CLINICAL TRIAL: NCT00823368
Title: Biomarker Testing and DNA Collection in Subjects Participating in a Double-Blind, Placebo-Controlled, Crossover, Flexible-Dose Evaluation of the Efficacy, Safety, and Tolerability of STX209 in the Treatment of Irritability in Subjects With Fragile X Syndrome
Brief Title: Biomarker Testing and DNA Collection in Subjects Participating in Protocol 22001
Status: Completed | Type: Observational
Sponsor: Seaside Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 22001A
Record Dates: First submitted 2009-01-13; First posted 2009-01-15 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-07

CONDITIONS: Fragile X Syndrome
Keywords: fragile X syndrome; biomarkers
MeSH Terms: conditions — Fragile X Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA from blood,plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Arbaclofen followed by Placebo
  Interventions: Drug: STX209
- Placebo followed by Arbaclofen
  Interventions: Drug: STX209

INTERVENTIONS:
Drug: STX209

SUMMARY:
The subjects that meet the inclusion and exclusion criteria and consent to participate in protocol 22001 will be offered participation in 22001A which will evaluate secreted protein before and after treatment with STX209 and placebo to determine if they correlate with effectiveness of treatment or susceptibility to treatment with STX209. These same subjects will also be asked to contribute a blood sample for DNA (deoxyribonucleic acid) collection. The investigators will study the DNA to determine if STX209 works better in people with specific gene variations, or to find new gene variations that predict how well STX209 works.

ELIGIBILITY:
Inclusion Criteria:

* Subjects that meet the inclusion and exclusion criteria and consent to participate in protocol 22001

Exclusion Criteria:

* Subjects that meet the inclusion and exclusion criteria and consent to participate in protocol 22001

Ages: 6 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Fragile x syndrome subjects that meet the inclusion and exclusion criteria and consent to participate in protocol 22001
Sampling Method: Non-Probability Sample
Dates: Start 2009-01; Primary Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
change in plasma proteins with treatment | After 4 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Berry-Kravis, MD, PhD, Principal Investigator — Rush University Medical Center; Randi Hagerman, MD, Principal Investigator — M.I.N.D. Institute; Craig Erikson, MD, Principal Investigator — Riley Hospital for Children; Bryan King, MD, PhD, Principal Investigator — Seattle Children's Hospital; James McCracken, MD, Principal Investigator — University of California, Los Angeles; Jonathan Picker, MBChB, PhD, Principal Investigator — Boston Children's Hospital; Linmarie Sikich, MD, Principal Investigator — University of North Carolina Neurosciences Hospital; Jeremy Veenstra-VanderWeele, MD, Principal Investigator — Vanderbilt Kennedy Center; Ted Brown, MD, PhD, Principal Investigator — NYS Institute for Basic Research in Developmental Disabilities; Lawrence Ginsberg, MD, Principal Investigator — Red Oaks Psychiatry Associates, PA; Shivkumar Hatti, MD, Principal Investigator — Suburban Research Associates; Raun Melmed, MD, Principal Investigator — Southwest Autism Research & Resource Center
Locations (11):
- United States (11):
  - Southwest Autism Research & Resource Center, Phoenix, Arizona
  - University of California-Los Angeles Neuropsychiatric Institute, Los Angeles, California
  - M.I.N.D. Institute, Sacramento, California
  - Rush University Medical Center, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - NYS Institute for Basic Research in Developmental Disabilities, Staten Island, New York
  - University of North Carolina Neurosciences Hospital, Chapel Hill, North Carolina
  - Suburban Research Associates, Media, Pennsylvania
  - Vanderbilt Kennedy Center, Nashville, Tennessee
  - Red Oaks Psychiatry Associates, PA, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington